CLINICAL TRIAL: NCT01999582
Title: A Phase 2 Multicenter, Randomized, Open-Label , Multiple-Dose Study of Intravenous and Subcutaneous Administration of Sotatercept (ACE-011) in Subjects With End-Stage Kidney Disease on Hemodialysis Switched From Erythropoeisis Stimulating Agents With Staggered Dose Group Escalation in Part 1 Followed by a Parallel Group, Active Controlled Study of Selected Dose(s) and Regimen(s) in Part 2: To Evaluate the Pharmacokinetics, Safety, Tolerability, Efficacy, Dosing Regimen, and Pharmacodynamics of Sotatercept
Brief Title: A Phase 2 Study of Intravenous or Subcutaneous Dosing of Sotatercept (ACE-011) in Patients With End-Stage Kidney Disease on Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-011-REN-002; 2012-003788-23 (EudraCT Number)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Anemia; Kidney Failure, Chronic
Keywords: Anemia; End Stage Kidney Disease; Chronic Kidney Disease; Dialysis; Erythrpoietin Stimulating Agent (ESA)
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Dose Group 1, 2, and 3 (Experimental): Intravenous Dose Group 1 starting at 0.1 mg/kg and escalated in Dose Groups 2 (0.2 mg/kg) and Dose Group 3 (0.1, 0.2, 0.3, 0.4 mg/kg, titrated based on titration rules, administered every 14 days)
  Interventions: Biological: Sotatercept
- Subcutaneous Dose Group 1, 2, and 3 (Experimental): Subcutaneous Dose Group 1 starting at 0.13 mg/kg and escalated in Dose Groups 2 (0.26 mg/kg) and Dose Group 3 (0.4 to 0.5 mg/kg, titrated based on titration rules, administered every14 days)
  Interventions: Biological: Sotatercept

INTERVENTIONS:
Biological: Sotatercept — Sotatercept is dosed intravenously every 14 days. The dose a subject receives will depend on the randomization arm and the dose group.
  Other Names: ACE-011
  Arms: Intravenous Dose Group 1, 2, and 3
Biological: Sotatercept — Sotatercept is dosed subcutaneously every 14 days. The dose a subject receives will depend on the randomization arm and the dose group.
  Other Names: ACE-011
  Arms: Subcutaneous Dose Group 1, 2, and 3

SUMMARY:
To determine the optimal route of administration, dose level, and safety of intravenous and subcutaneous dosing of sotatercept for maintaining hemoglobin levels in subjects who are on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age.
2. Subjects on at least 6 hours of hemodialysis per week, for at least 12 weeks before screening
3. Subjects must be on a stable intravenous or subcutaneous dose of Erythropoietin Stimulating Agents (excluding methoxy polyethylene glycol-epoetin beta [Mircera]) to maintain hemoglobin.
4. A mean predialysis hemoglobin concentration ≥ 10 g/dL (grams per deciliter) to ≤ 12 g/dL (≥ 100 g/L (grams per liter) to ≤ 120 g/L) obtained from three consecutive days.

4. A Body Mass Index value ≥ 18.5 kg/m2 (kilograms per m2) at screening. 5. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.

6. Able to adhere to the study visit schedule and comply with all protocol requirements.

Exclusion Criteria:

1. Non renal causes of anemia
2. Subjects on peritoneal dialysis.
3. Systemic hematological disease
4. Uncontrolled diabetes mellitus (HbA1c (hemoglobin A1c) > 9%) at screening.
5. Uncontrolled hypertension defined as mean of home systolic blood pressure > 160 mm Hg (millimeter of mercury) or mean of home diastolic blood pressure > 90 mm Hg calculated once during the screening period prior to randomization
6. Subjects with heart failure
7. History of malignancy (except excised and cured non-melanoma skin cancer, or cervical carcinoma in situ that was surgically ablated more than 5 years ago).
8. Anticipated or scheduled living donor renal transplant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11-30 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Smith, MD, Study Director — Celgene Corporation
Locations (23):
- Belgium (3):
  - Centre Hospitalier EpiCURA - Clinique Louis Caty de Baudour, Baudour
  - Universitaire Ziekenhuizen (UZ) Leuven - Gasthuisberg, Leuven
  - CHR de la CITADELLE, Liège
- Germany (4):
  - KfH Nierenzentrum Coburg, Coburg
  - Gemeinschaftspraxis und Dialysezentrum Karlstrass, Düsseldorf
  - KfH Kuratorium für Dialyse und Nierentransplantation e.v., München
  - KfH Nierenzentrum Rosenheim, Rosenheim
- Portugal (3):
  - Nephrocare Faro, Faro
  - Hospital de Santa Maria, Lisbon
  - Nephrocare Portimao, Portimão
- Spain (10):
  - Complejo Hospitalario de Torrecardenas, Almería
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Galdakao-Usansolo, Galdakao
  - Servicio de Nefrologia Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital de Torrevieja, Torrevieja (Alicante)
- United Kingdom (3):
  - Cambridge University Hospitals NHS Trust, Cambridge
  - Glasgow Royal Infirmary, Glasgow
  - St Georges Healthcare NHS Trust, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection: Participants received sotatercept at 0.1 mg/kg administered IV every 14 days for up to 8 doses to evaluate the Pharmacokinetic (PK) and safety of IV versus subcutaneous (SQ) dosing of sotatercept.
- Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection: Participants received sotatercept at 0.13 mg/kg administered SC every 14 days for up to 8 doses to evaluate the PK and safety of IV versus SC dosing of sotatercept.
- Group 2: Sotatercept 0.2 mg/kg IV Injection: Participants received sotatercept at 0.2 mg/kg administered IV every 14 days for up to 8 doses to evaluate the PK and safety of IV versus SC dosing of sotatercept.
- Group 2: Sotatercept 0.26 mg/kg SC Injection: Participants received sotatercept at 0.26 mg/kg administered SC every 14 days for up to 8 doses to evaluate the PK and safety of IV versus SC dosing of sotatercept.
- Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection: Participants received sotatercept at a starting dose of 0.1 mg/kg. Intra subject dose escalation will be implemented in response to subjects' individual hemoglobin levels and can be increased in 0.1 mg/kg increments up to 0.4 mg/kg administered IV every 14 days for up to 8 doses to evaluate the PK and safety of IV versus SC dosing of sotatercept.
- Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection: Participants received sotatercept at 0.4 mg/kg. Intra subject dose escalation will be implemented in response to subjects' individual hemoglobin levels and can be increased in 0.1 mg/kg increments up to 0.5 mg/kg administered SC every 14 days for up to 8 doses to evaluate the PK and safety of IV versus SC dosing of sotatercept.
Period: Overall Study
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Started | 7 | 7 | 9 | 9 | 12 | 6
Completed | 4 | 4 | 3 | 6 | 10 | 3
Not Completed | 3 | 3 | 6 | 3 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 1 | 0
Not completed — Other Reasons | 1 | 0 | 3 | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 3 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection | Total
Number analyzed (Participants) | 7 | 7 | 9 | 9 | 12 | 6 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (15.43) | 62.3 (13.03) | 59.4 (15.8) | 61.9 (15.43) | 61.4 (15.68) | 53.7 (15.93) | 60.0 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 3 | 5 | 3 | 22
  Male | 3 | 4 | 5 | 6 | 7 | 3 | 28
Race [Count of Participants; unit: Participants]
  White | 4 | 5 | 6 | 8 | 11 | 6 | 40
  Black or African- American | 1 | 1 | 1 | 0 | 1 | 0 | 4
  Asian | 2 | 0 | 2 | 1 | 0 | 0 | 5
  American Indian/Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 7 | 6 | 8 | 9 | 12 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-Time Curve Over Dosing Interval (AUC14d) (14 Days)
Description: Area Under the plasma concentration-time curve over 14-day dosing interval (AUC14) for Sotatercept., The PK population included all participants in the safety population with at least one non-missing plasma concentration data. All analyses of PK data were based on the PK population and participants were analyzed according to the treatment group to which they were randomized.
Time Frame: Doses 1-2: predose and postdose at 5 min (IV only) 4 hours, 3, and 7 days after each dose; Doses 3-7: predose, and postdose at 5 min after IV injection after each dose; Final dose: predose and postdose at 5 min (IV only) 4 hours, 3, 7, 14 days after dose
Population: Pharmacokinetic population-all treated participants with at least one non-missing plasma concentration data for this endpoint
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 7 | 5
day*ng/mL | 15204.31 (7096.55) [lower limit 7096.55] | 11269.14 (1839.92) [lower limit 1839.92] | 28647.03 (10332.19) [lower limit 10332.19] | 10327.98 (8065.12) [lower limit 8065.12] | 15886.83 (4212.12) [lower limit 4212.12] | 21982.9 (5125.4) [lower limit 5125.4]

2. Primary Outcome: Area Under the Serum Concentration- Time Curve Over From Day 1 to Day 28 (AUC28d)
Description: Area under the plasma concentration-time curve over 28-day dosing interval (AUC28d). All analyses of PK data were based on the PK population and participants were analyzed according to the treatment group to which they were randomized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 5 | 2
day*ng/mL | 38361.5 (8589.34) [lower limit 8589.34] | 41500.36 (13647.28) [lower limit 13647.28] | 94106.54 (37204.17) [lower limit 37204.17] | 36065.09 (22817) [lower limit 22817] | 33173.4 (8709.16) [lower limit 8709.16] | 60497.8 (14623.13) [lower limit 14623.13]

3. Primary Outcome: Maximum Observed Serum Concentration Obtained From the First Dose (Cmax14d)
Description: Maximum observed serum concentration (Cmax14d) of sotatercept, obtained directly from the observed concentration-time data. The PK population included all participants in the safety population with at least one non-missing plasma concentration data. All analyses of PK data were based on the PK population and participants were analyzed according to the treatment group to which they were randomized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 4 | 3 | 8 | 6 | 7 | 5
ng/mL | 2567.6 (1093.73) [lower limit 1093.73] | 1024.27 (145.8) [lower limit 145.8] | 4623.61 (1620.66) [lower limit 1620.66] | 963.05 (659.65) [lower limit 659.65] | 3155.53 (1861.07) [lower limit 1861.07] | 1993.58 (375.54) [lower limit 375.54]

4. Primary Outcome: Maximum Observed Serum Concentration (Cmax28d) Obtained From the Combined First 2 Doses
Description: Maximum observed serum concentration (Cmax28d) of sotatercept, obtained directly from the observed concentration-time data combining the profiles following the first two doses. The PK population included all participants in the safety population with at least one non-missing plasma concentration data. All analyses of PK data were based on the PK population and participants were analyzed according to the treatment group to which they were randomized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 5 | 2
ng/mL | 3557.93 (699.19) [lower limit 699.19] | 3868.83 (3614.89) [lower limit 3614.89] | 8613.67 (3559.69) [lower limit 3559.69] | 1967.55 (1128.69) [lower limit 1128.69] | 3501.54 (2144.15) [lower limit 2144.15] | 3161.6 (788.14) [lower limit 788.14]

5. Primary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax)
Description: Time to maximum serum concentration (Tmax) of sotatercept, obtained directly from the observed concentration-time data. The PK population included all participants in the safety population with at least one non-missing plasma concentration data. All analyses of PK data were based on the PK population and participants were analyzed according to the treatment group to which they were randomized.
Time Frame: Doses 1-2: pre- and postdose at 5 min (IV only) 4 hrs, 3, and 7 days after each dose; Doses 3-7: pre-, and postdose at 5 min after IV injection after each dose; Final dose: pre- and postdose at 5 min (IV only), 4 hrs, 3, 7, 14, 28, 56, 84, and 112 days
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 4 | 3 | 3 | 4 | 5 | 2
days | 14.09 (14.01) [14.01 to 16] | 21.01 (16.16) [16.16 to 27.98] | 14.02 (13.99) [13.99 to 16.01] | 18.51 (15.99) [15.99 to 21.02] | 0.1688 (0.0035) [0.0035 to 15.99] | 21.06 (20.99) [20.99 to 21.13]

6. Primary Outcome: Estimate of Terminal Elimination Half-Life in Serum at Final Dose Only (t1/2)
Description: Terminal elimination half-life (T1/2). The PK population included all participants in the safety population with at least one non-missing plasma concentration data. All analyses of PK data were based on the PK population and participants were analyzed according to the treatment group to which they were randomized.
Time Frame: Predose and postdose at 5 min (IV only) 4 hours, 3, 7, 14, 28, 56, 84, and 112 days after the final dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 6 | 4 | 6 | 8 | 9 | 4
days | 17.6 (4.631) [lower limit 4.631] | 25.87 (7.127) [lower limit 7.127] | 21.76 (3.941) [lower limit 3.941] | 21.03 (5.4) [lower limit 5.4] | 22.46 (5.342) [lower limit 5.342] | 20.39 (5.3) [lower limit 5.3]

7. Primary Outcome: Lambda (ʎz): Apparent Terminal Rate Constant (at Final Dose Only)
Description: Lambda, apparent terminal rate constant (final dose only). The PK population included all participants in the safety population with at least one non-missing plasma concentration data. All analysis of PK data were based on the PK population and participants were analyzed according to the treatment group to which they were randomized.
Time Frame: Predose and postdose at 5 min (IV only) 4 hours, 3, 7, 14, 28, 56, 84, and 112 days after the final dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/day
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 6 | 4 | 6 | 8 | 4 | 4
1/day | 0.0414 (0.0094) [lower limit 0.0094] | 0.0282 (0.0071) [lower limit 0.0071] | 0.0328 (0.0063) [lower limit 0.0063] | 0.0346 (0.0078) [lower limit 0.0078] | 0.0326 (0.0085) [lower limit 0.0085] | 0.0355 (0.0077) [lower limit 0.0077]

8. Secondary Outcome: Percentage of Participants With Mean Hemoglobin ≥ 100 g/L to ≤ 120 g/L Without Rescue Medication
Description: The percentage of participants able to maintain a mean (Visit 14 to 17) hemoglobin concentration ≥ 100 g/L to ≤ 120 g/L without the need for rescue medication at each dose level. Mean hemoglobin value is a mean of hemoglobin concentrations from Visit 14 to Visit 17 (days 99 to 113).
Time Frame: Visit 14 to Visit 17 (days 99 to 113)
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 7 | 7 | 9 | 9 | 12 | 6
Percentage of participants | 42.9 | 42.9 | 11.1 | 33.3 | 25 | 50

9. Secondary Outcome: Change From Baseline in Mean Hemoglobin Concentration for Visit 14 to 17 (All Participants Regardless of Rescue)
Description: Change in mean hemoglobin concentration between baseline and Visit 14 to 17 at each dose level. Baseline hemoglobin value is the mean of three consecutive hemoglobin concentrations with the last hemoglobin concentration done within the 7 days prior to randomization and the value obtained on the day of randomization. Visit 14 to 17 hemoglobin value is a mean of hemoglobin concentrations from Day 99 [Visit 14] to Day 113 [Visit 17].
Time Frame: Baseline and Visit 14 to Visit 17 (days 99 to 113)
Population: All randomized participants who received at least one dose of treatment.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 7 | 5 | 5 | 7 | 9 | 4
g/L | -6.9 (11.61) [lower limit 11.61] | -2.7 (6.47) [lower limit 6.47] | -2.1 (12.23) [lower limit 12.23] | -0.8 (10.03) [lower limit 10.03] | -9.9 (9.3) [lower limit 9.3] | -6.4 (12.6) [lower limit 12.6]

10. Secondary Outcome: Change From Baseline in Mean Hemoglobin Concentration for Visit 14 to 17 (Participants Not Rescued Prior to Day 115)
Description: Change in mean hemoglobin concentration between baseline and Visit 14 to 17 at each dose level for participants not rescued prior to Day 115. Baseline hemoglobin value is the mean of three consecutive hemoglobin concentrations with the last hemoglobin concentration done within the 7 days prior to randomization and the value obtained on the day of randomization. Visit 14 to 17 hemoglobin value is a mean of hemoglobin concentrations from Day 99 [Visit 14] to Day 113 [Visit 17].
Time Frame: Baseline and Visit 14 to Visit 17 (days 99 to 113)
Population: All randomized participants who received at least one dose of treatment and were not rescued prior to Day 115.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 3 | 4 | 2 | 6 | 6 | 3
g/L | -7 (6.24) [lower limit 6.24] | -3.6 (7.08) [lower limit 7.08] | -0.3 (15.2) [lower limit 15.2] | 0.5 (10.28) [lower limit 10.28] | -13 (10.07) [lower limit 10.07] | -1 (8.05) [lower limit 8.05]

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Treatment-emergent adverse event (TEAE) was defined as an adverse event with start date on or after date of first dose of study drug. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participants during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. A serious adverse event is defined as any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. Severity and intensity was assessed using the following grading scale: Mild, Moderate and Severe (could be non-serious or serious).
Time Frame: From date of first dose of investigational product to 112 days after the last dose or until the last study visit, whichever period was longer. The maximum duration for any IV or SC dose was 114 days. Up to approximately 226 days.
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
Number analyzed (Participants) | 7 | 7 | 9 | 9 | 12 | 6
Participants
  Any TEAE | 7 | 3 | 9 | 6 | 10 | 6
  Any Treatment-Related TEAE | 1 | 1 | 1 | 0 | 0 | 1
  Any Serious TEAE | 3 | 0 | 3 | 1 | 3 | 3
  Any Treatment-Related Serious TEAE | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to study drug discontinuation | 0 | 0 | 3 | 0 | 1 | 0
  Any Severe TEAE | 0 | 0 | 2 | 0 | 1 | 2
  Any TEAE Leading to Death | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of first dose to study completion (up to approximately 33 months). Serious Adverse events and other adverse events were assessed from date of first dose to 112 days after the last dose or until the last study visit, whichever period was longer, up to approximately 226 days.
Arm/Group | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection | Group 2: Sotatercept 0.2 mg/kg IV Injection | Group 2: Sotatercept 0.26 mg/kg SC Injection | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/9 | 0/9 | 0/12 | 1/6
Serious Adverse Events (participants affected / at risk) | 3/7 | 0/7 | 3/9 | 1/9 | 3/12 | 3/6
Other Adverse Events (participants affected / at risk) | 7/7 | 3/7 | 9/9 | 6/9 | 9/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection (N=7) | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection (N=7) | Group 2: Sotatercept 0.2 mg/kg IV Injection (N=9) | Group 2: Sotatercept 0.26 mg/kg SC Injection (N=9) | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection (N=12) | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection (N=6)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Sotatercept 0.1 mg/kg Intravenous (IV) Injection (N=7) | Group 1: Sotatercept 0.13 mg/kg Subcutaneous (SC) Injection (N=7) | Group 2: Sotatercept 0.2 mg/kg IV Injection (N=9) | Group 2: Sotatercept 0.26 mg/kg SC Injection (N=9) | Group 3: Sotatercept 0.1 - 0.4 mg/kg IV Injection (N=12) | Group 3: Sotatercept 0.4 - 0.5 mg/kg SC Injection (N=6)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amaurosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choroidal effusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardioactive drug level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extravasation blood (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 1 (2) | 1 (3) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to a shift in the clinical development strategy for the renal sotatercept program, Part 2 of the study was not conducted; Part 2 objectives were not assessed and none of the statistical analyses in Part 2 were conducted; no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.